CLINICAL TRIAL: NCT07095387
Title: Eco-anxiety and Coping in Children: Results From a Pilot Randomized Cluster Trial Evaluating the Impact of a Creative Arts and Philosophical Inquiry Intervention for Elementary School Students
Brief Title: Pilot Study of a School Based Intervention for Coping With Climate Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Bishop's University (Other)
Responsible Party: Principal Investigator, Terra Léger-Goodes, Principal investigator, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 767-2023-1376; 767-2023-1376 (Other Grant/Funding Number: Social Science and Humanities Research Council of Canada (SSHRC))
Record Dates: First submitted 2025-07-01; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Eco-anxiety
Keywords: art-intervention; philosophy inquiry; eco-anxiety; coping with climate change; school-based intervention

STUDY DESIGN:
Intervention Model Description: Randomized cluster trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative arts an philosophy inquiry intervention (Experimental): The intervention group received the one workshop per week for 7 weeks. Each workshop combined artistic creation and group philosophical inquiry on a certain theme related to climate change (e.g., responsibility, hope, the beauty of nature)
  Interventions: Behavioral: Making room for climate emotions in the classroom
- Wait-list control group (No Intervention)

INTERVENTIONS:
Behavioral: Making room for climate emotions in the classroom — This intervention combined creative arts workshops using drawing, photography, painting and collage to introduce a theme related to climate change and promote emotional expression. The artistic creation was followed by a philosophical inquiry group discussion on a theme related to the artistic creation to allow critical thinking and sharing perceptions.
  Arms: Creative arts an philosophy inquiry intervention

SUMMARY:
The present study aimed to evaluate the impacts of a school-based program that combined creative arts and philosophy inquiry to discuss climate change emotions with children. The objective was to determine if there were changes that could be seen in the group that participated in the weekly workshops (total of 7 workshops) compared to the group who did not participate (control group). A questionnaire was administered to all children before the intervention began and after it finished to compare scores on the variables of coping with climate change, eco-anxiety, intolerance to distress, general anxiety, and self-determination.

ELIGIBILITY:
Inclusion Criteria:

* Elementary school student in recruited classrooms

Exclusion Criteria:

-

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Coping with climate change | Baseline and 8 weeks
  The Coping with Climate Change Scale for Adolescents developed by Ojala (2012) uses a Likert-type scale (0 = not true at all for me; 4 = completely true for me) to measure three coping dimensions (problem coping, avoidance coping, and meaning coping). Lower scores represent less usage of this coping strategy, while higher scores indicate high usage of this coping strategy.
Eco-anxiety | Baseline and 8 weeks
  The Hogg Eco-anxiety Scale (2021) was adapted to children by making the language more accessible. The scale is rated on a 4-point Likert type scale (0 = Never, 3 = Almost every day), and higher scores indicate higher eco-anxiety (worst outcomes).

SECONDARY OUTCOMES:
Intolerance to distress | Baseline and 8 weeks
  The Distress Intolerance Index for Youth (Keller, 2019) uses a 5-point Likert type scale (0 = Not at all true for me to 4 = Very true for me), and higher scores indicate higher intolerance to distress (worst outcome).
General anxiety | Baseline and 8 weeks
  The Behavior Assessment Scale for Children 3rd edition for Canadian francophones (BASC-III; Reynolds & Kamphaus, 2015) uses a Likert-type scale (0 = never to 3 = almost always), and higher scores indicate higher anxiety symptoms (worst outcome).
Self-determination | Baseline and 8 weeks
  The Self-Determination at School Scale (Savard et al., 2013) uses a 5-point Likert-type scale (from 0 = Almost never to 4 = Almost always) where higher scores indicate higher levels of self-determination (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Bishop's University, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) collected in this study will not be made publicly available, but can be obtained by contacting the researchers directly.